CLINICAL TRIAL: NCT01332032
Title: Promoting Breast Cancer Screening in Non-adherent Women
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Reliant Medical Group (Other); Fallon Community Health Plan (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary E. Costanza, Study Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: FCM001; R01CA132935 (NIH)
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: cost effectiveness; screening mammography; repeat mammography; telephone counseling; computerized reminders; compliance
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Reminder Letter: A letter sent to women reminding them that are coming due or overdue for a mammogram. It contains a reminder that their primary care provider (PCP) recommends mammography screening every 1-2 years. It urges them to call a special number to a study scheduler to get assistance scheduling a mammogram and is signed electronically by their primary care provider. Repeat "Booster" letters will be sent in subsequent years to those failing to get a mammogram.
  Interventions: Behavioral: Reminder Letter
- Reminder Call: A reminder letter (as in the 1st group) is sent. If a woman does not call in to schedule a mammogram within 2 weeks, a study scheduler will call her, remind her she is coming or is overdue, remind her that her PCP recommends screening every 1-2 years and offer to schedule a mammogram for her. Repeat "Booster" letters will be sent and repeat scheduler calls made in subsequent years to those failing to get a mammogram.
  Interventions: Behavioral: Reminder Call
- Counselor Call: A reminder letter as above is sent first. If a woman does not call in to schedule a mammogram within 2 weeks, a second letter is sent along with a mammography educational booklet. The second letter also reiterates a reminder that her PCP recommends screening every 1-2 years, and offers a special number to call to schedule. If a woman does not schedule within 8-10 days, a counselor will call. The protocol script included tailored barriers counseling, correction of misinformation and motivational interviewing. Repeat "booster" letters will be sent and repeat counselors calls made in subsequent years to those failing to get a mammogram. techniques. Average calls last 20-30 minutes.
  Interventions: Behavioral: Counselor Call

INTERVENTIONS:
Behavioral: Reminder Letter — A letter sent to women reminding them that they are coming due or overdue for a mammogram. It contains a reminder that their doctor recommends mammography screening every 1-2 years; urges them to call a special number to a study scheduler to get assistance scheduling a mammogram and is signed electronically by their primary care provider. For women in the reminder letter only arm, who did not complete a mammogram within 12 months of the first reminder, a booster intervention (I.E. reminder letter) will be sent. The letter requests that a woman call in to schedule a mammogram, and reminds her that her PCP recommends she get one. Booster letters will be sent up to three times at annual intervals for those failing to get a mammogram
  Other Names: mammography reminder letter.
  Groups: Reminder Letter
Behavioral: Reminder Call — A reminder letter (as in the 1st group) is sent. If a woman does not call in to schedule a letter, 2 weeks later, a study scheduler will call her, remind her she is coming or is overdue, remind her that her PCP recommends screening every 1-2 years and offers to schedule a mammogram for her. For women in the reminder letter arm who did not complete a mammogram within 12 months of the first reminder, a booster intervention ( I.E.a reminder letter will be sent requesting that they call in to schedule a mammogram. The letter reminds her that her PCP recommends she get a mammogram. Those who do not respond within 7 days, will receive a scheduler call) will be repeated as necessary for up to 3 times.
  Other Names: mammography phone call
  Groups: Reminder Call
Behavioral: Counselor Call — Reminder letter s as above is sent. If subject does not call in to schedule within 2 weeks, second letter is sent with mammography educational booklet. Second letter reiterates reminder that PCP recommends screening. Has number to call to schedule. If subject does not schedule within 2 weeks, counselor will call. Protocol script includes tailored barriers counseling, correction of misinformation and motivational interviewing techniques. For those who did not complete a mammogram within 12 months of the first reminder, a booster intervention will be repeated annually for up to 3 times as necessary.Booster is reminder letter with pamphlet stressing the 4 reasons why women need regular mammograms.
  Other Names: educator call
  Groups: Counselor Call

SUMMARY:
This randomized study compares the effectiveness and cost-effectiveness of 3 proven methods of reaching out to women who are coming due for or who are overdue for a mammogram. The study originally embedded in a community healthcare plan and an associated community clinic, now accepts patients using the community clinic and 3 other health care plans. The study makes use of a complex computer driven reminder system.

The study also will examine ways to improve the efficiency and sequencing of the interventions by identifying patient factors associated with intervention effectiveness.

DETAILED DESCRIPTION:
The randomized study compares three interventions. All eligible women are randomly assigned to 1 of 3 interventions. If they become 18 or more months from a prior mammogram, they will receive the intervention to which they were assigned.

The 3 arms are

1. RL ARM: (reminder letter) a control arm which consists of a reminder letter only that states when the last mammogram was, contains a standard recommendation from her primary care provider (PCP), and requests that the woman call a special number for help scheduling a mammogram.
2. RC ARM: (reminder call) a reminder letter as above, followed, if no response, by a reminder call from a study scheduler who offers to help schedule a mammogram.
3. ETTC ARM: (enhanced tailored telephone counseling call) a reminder letter as above, followed, if no response by a second letter, a mammography educational booklet and a second request to call a special number to schedule a mammogram. If no response, a study counselor/educator will call.

A complex computer-based tracking system identifies women coming due for a mammogram or those overdue for a mammogram. The system interfaces with the clinic database systems and stores information re age, telephone number, address, prior screening dates, primary care provider name, scheduling dates, etc. The system can generate reminder letters as appropriate.

The tracking system also interfaces with computer-assisted telephone script systems(CATI) which prompt the study scheduler or the study counselor to follow the protocol that is tailored to the individual patient.

The CATI system captures data from all calls, including how ready a woman is to schedule, the answers to a brief socio-demographic survey and in the counselor call script barriers and misinformation about mammography.

The computer system also interfaces with the radiology scheduling system so that study personnel can assist women in scheduling a mammogram during the phone call.

The primary outcome is the number of women in each arm getting a mammogram. This data will come from the clinic data base and the healthcare plan billing system.

Secondary outcomes include evaluation of the effect of booster or repeat interventions in women failing to respond to prior request for mammogram.

ELIGIBILITY:
Inclusion Criteria:

* women aged 40 through 84 years old
* in the Fallon Community Health Plan, Blue Cross, Tufts or Harvard Pilgrim health plans for 18 or more months
* has a current Reliant Medical Group (formerly called Fallon Clinic) primary care provider
* has working telephone

Exclusion Criteria:

* significant cognitive impairment
* serious illness, precluding screening
* bilateral mastectomy
* life expectancy less than 5 years

Ages: 40 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 40 to 84 who have life expectancy of five years, have at least one breast, and who have been cared for by Fallon Community Health Plan and currently cared for by Reliant Medical Group (formerly called Fallon Clinic) PCP. Interventions directed at women who are at least 18 months from prior mammogram. Since July 2012, patients with a current Reliant Medical Group PCP who have been enrolled in Blue Cross/Bluse Shield, Harvard Pilgrim or Tufts health plans for 18 months may be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 36348 (Actual)
Dates: Start 2009-07; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The proportion of women in each arm who complete a mammogram in the prior 24 months | 4 years
  The outcome will be determined for each of the 4 years of intervention. But the main interest will be the outcome measured in the final intervention year because we believe this best illustrates the magnitude of intervention effect that could be achieved in future years.

SECONDARY OUTCOMES:
A comparison of the number of interventions required per arm | 4 years
  We anticipate that fewer women who receive the ETTC call (Counselor call) will need repeat interventions compared with the women in the reminder call arm or the women in the reminder letter arm.
The percent of women in each arm receiving an intervention who will complete a scheduled mammogram | 4 years
  We anticipate that women who received a counselor (ETTC) call and who scheduled a mammogram on the call will have the highest completion rate compared to women who received a reminder call or a reminder letter.
Evaluation of the effectiveness of booster or repeat interventions in women failing to respond to request for getting a mammogram | 4 years
  The relative effectiveness and cost effectiveness of repeating reminders (letters, calls vs. counseling calls) in women who have not responded to a prior request(s) for completing a mammogram will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Costanza, MD, Principal Investigator — UMass Medical School and Reliant Medical Group (formerly called Fallon Clinic); Roger Luckmann, MD, MPH, Principal Investigator — UMass Medical School
Locations (1):
- Reliant Medical Group, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Costanza ME, Luckmann R, White MJ, Rosal MC, Cranos C, Reed G, Clark R, Sama S, Yood R. Design and methods for a randomized clinical trial comparing three outreach efforts to improve screening mammography adherence. BMC Health Serv Res. 2011 Jun 3;11:145. doi: 10.1186/1472-6963-11-145. PMID 21639900